CLINICAL TRIAL: NCT03285711
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study Evaluating the Safety and Efficacy of Filgotinib and GS-9876 in Subjects With Lupus Membranous Nephropathy (LMN)
Brief Title: Study to Evaluate the Safety and Efficacy of Filgotinib and Lanraplenib in Adults With Lupus Membranous Nephropathy (LMN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-437-4093
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Lupus Membranous Nephropathy
MeSH Terms: interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lanraplenib 30 mg (Experimental): Participants receive lanraplenib 30 mg tablet + filgotinib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase. Participants who achieve ≥ 35% reduction in urinary protein excretion from baseline continue to receive same blinded study treatment for additional 16 weeks. Participants who did not achieve a ≥ 35% reduction in urinary protein excretion will switch treatment.
  After 32 weeks of blinded treatment, participants who have ≥ 35% reduction in urinary protein excretion from baseline continue their assigned blinded treatment for additional 20 weeks in Extended Blinded Treatment Phase.
  Interventions: Drug: Lanraplenib; Drug: Filgotinib placebo
- Filgotinib 200 mg (Experimental): Participants receive filgotinib 200 mg tablet + lanraplenib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase. Participants who achieve ≥ 35% reduction in urinary protein excretion from baseline continue to receive same blinded study treatment for additional 16 weeks. Participants who did not achieve a ≥ 35% reduction in urinary protein excretion will switch treatment.
  After 32 weeks of blinded treatment, participants who have ≥ 35% reduction in urinary protein excretion from baseline continue their assigned blinded treatment for additional 20 weeks in Extended Blinded Treatment Phase.
  Interventions: Drug: Filgotinib; Drug: Lanraplenib placebo
- Lanraplenib 30 mg to Filgotinib 200 mg (Experimental): At Week 16, participants who do not achieve a ≥ 35% reduction in urinary protein excretion from baseline to Week 16 switch treatment and receive filgotinib 200 mg + lanraplenib placebo for additional 16 weeks.
  At Week 32, participants who do not achieve a ≥ 35% reduction in urinary protein excretion from Week 16 to Week 32 can continue whichever treatment that lead to the greatest reduction in urinary protein excretion, or either treatment per investigator's discretion for additional 20 weeks in Extended Blinded Treatment Phase.
  Interventions: Drug: Filgotinib; Drug: Lanraplenib placebo
- Filgotinib 200 mg to Lanraplenib 30 mg (Experimental): At Week 16, participants who do not achieve a ≥ 35% reduction in urinary protein excretion from baseline to Week 16 switch treatment and receive lanraplenib 30 mg + filgotinib placebo for additional 16 weeks.
  At Week 32, participants who do not achieve a ≥ 35% reduction in urinary protein excretion from Week 16 to Week 32 can continue whichever treatment that lead to the greatest reduction in urinary protein excretion, or either treatment per investigator's discretion for additional 20 weeks in Extended Blinded Treatment Phase.
  Interventions: Drug: Lanraplenib; Drug: Filgotinib placebo

INTERVENTIONS:
Drug: Filgotinib — 200 mg tablet administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 200 mg; Lanraplenib 30 mg to Filgotinib 200 mg
Drug: Lanraplenib — 30 mg tablet administered orally once daily
  Other Names: GS-9876
  Arms: Filgotinib 200 mg to Lanraplenib 30 mg; Lanraplenib 30 mg
Drug: Filgotinib placebo — Tablet administered orally once daily
  Arms: Filgotinib 200 mg to Lanraplenib 30 mg; Lanraplenib 30 mg
Drug: Lanraplenib placebo — Tablet administered orally once daily
  Arms: Filgotinib 200 mg; Lanraplenib 30 mg to Filgotinib 200 mg

SUMMARY:
The primary objective of this study is to evaluate the efficacy of filgotinib and lanraplenib (previously GS-9876) in adults with lupus membranous nephropathy (LMN).

ELIGIBILITY:
Key Inclusion Criteria:

* Kidney biopsy within the 36 months prior to screening with a histologic diagnosis of LMN (International Society of Nephrology [ISN] and the Renal Pathology Society [RPS] 2003 classification of lupus nephritis), either Class V alone, or Class V in combination with Class II.
* Urine protein excretion ≥ 1.5 grams per day
* Estimated glomerular filtration rate (eGFR) ≥ 40 mg/min/1.73m^2 based on the modification of diet in renal disease (MDRD) formulation at screening
* No evidence of active or latent tuberculosis (TB) as assessed during screening

Key Exclusion Criteria:

* Prior treatments as follows:

  * Previous treatment with a janus kinase (JAK) inhibitor within 3 months of Day 1
  * Use of rituximab or other selective B lymphocyte depleting agents (including experimental agents) within 6 months of Day 1. Enrollment is permitted if the last dose was given > 6 months and CD19-positive B cells are detectable at Screening.
* Use of any concomitant prohibited medications as described in the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2020-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Monitor, Study Director — Gilead Sciences
Locations (7):
- United States (7):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of Florida, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina at Chapel Hill / UNC School of Medicine, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baker M, Chaichian Y, Genovese M, Derebail V, Rao P, Chatham W, Bubb M, Lim S, Hajian H, Gurtovaya O, Patel U, Tumlin J. Phase II, randomised, double-blind, multicentre study evaluating the safety and efficacy of filgotinib and lanraplenib in patients with lupus membranous nephropathy. RMD Open. 2020 Dec;6(3):e001490. doi: 10.1136/rmdopen-2020-001490. PMID 33380521

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 06 October 2017. The last study visit occurred on 03 February 2020.
Pre-assignment Details: 22 participants were screened.
Groups:
- Lanraplenib 30 mg: Participants received lanraplenib 30 mg tablet + filgotinib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase. Participants who achieved ≥ 35% reduction in urinary protein excretion from baseline continued to receive same blinded study treatment for additional 16 weeks.
  After 32 weeks of blinded treatment, participants who had ≥ 35% reduction in urinary protein excretion from baseline continued their assigned blinded treatment for additional 20 weeks in Extended Blinded Treatment Phase.
- Filgotinib 200 mg: Participants received filgotinib 200 mg tablet + lanraplenib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase. Participants who achieved ≥ 35% reduction in urinary protein excretion from baseline continued to receive same blinded study treatment for additional 16 weeks.
  After 32 weeks of blinded treatment, participants who had ≥ 35% reduction in urinary protein excretion from baseline continued their assigned blinded treatment for additional 20 weeks in Extended Blinded Treatment Phase.
- Lanraplenib 30 mg to Filgotinib 200 mg: At Week 16, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from baseline to Week 16 switched treatment and received filgotinib 200 mg + lanraplenib placebo for additional 16 weeks.
  At Week 32, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from Week 16 to Week 32 could continue whichever treatment that led to the greatest reduction in urinary protein excretion, or either treatment per investigator's discretion for additional 20 weeks in Extended Blinded Treatment Phase.
- Filgotinib 200 mg to Lanraplenib 30 mg: At Week 16, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from baseline to Week 16 switched treatment and received lanraplenib 30 mg + filgotinib placebo for additional 16 weeks.
  At Week 32, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from Week 16 to Week 32 could continue whichever treatment that led to the greatest reduction in urinary protein excretion, or either treatment per investigator's discretion for additional 20 weeks in Extended Blinded Treatment Phase.
Period: Blinded Phase (Up to Week 16)
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Lanraplenib 30 mg to Filgotinib 200 mg | Filgotinib 200 mg to Lanraplenib 30 mg
Started | 4 | 5 | 0 | 0
Completed | 1 | 4 | 0 | 0
Not Completed | 3 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Period: Blinded Phase (Week 16 to 32)
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Lanraplenib 30 mg to Filgotinib 200 mg | Filgotinib 200 mg to Lanraplenib 30 mg
Started | 0 (1 participant switched treatment to filgotinib.) | 3 (1 participant switched treatment to lanraplenib.) | 1 (1 participant switched treatment from lanraplenib.) | 1 (1 participant switched treatment from filgotinib.)
Completed | 0 | 3 | 0 | 1
Not Completed | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Period: Extended Blinded Phase (Week 32 to 52)
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Lanraplenib 30 mg to Filgotinib 200 mg | Filgotinib 200 mg to Lanraplenib 30 mg
Started | 0 | 3 | 0 | 1
Completed | 0 | 2 | 0 | 1
Not Completed | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Lanraplenib 30 mg: Participants were randomized to receive lanraplenib 30 mg tablet + filgotinib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase.
- Filgotinib 200 mg: Participants were randomized to receive filgotinib 200 mg tablet + lanraplenib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase.
- Total: Total of all reporting groups
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (15.8) | 35 (16.9) | 35 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
24-Hour Urine Protein [Mean (Standard Deviation); unit: g/day] | 6.0 (4.65) | 3.3 (2.47) | 4.5 (3.62)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 116.1 (55.41) | 102.6 (30.61) | 108.6 (40.87)
Urine Protein Creatinine Ratio (UPCR) [Mean (Standard Deviation); unit: mg/mg] | 5.1 (4.38) | 1.9 (1.04) | 3.3 (3.23)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Urine Protein From Baseline (Day 1) to Week 16
Description: Urine protein was assessed by urinary protein excretion during a 24-hour urine collection.
Time Frame: Baseline; Week 16
Population: Participants in the Full Analysis Set (included all randomized participants who took at least 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 1 | 4
percent change | -2.8 | -51.2 (25.67)

2. Secondary Outcome: Change From Baseline (Day 1) in Urine Protein at Week 16
Description: Urine protein was assessed by urinary protein excretion during a 24-hour urine collection.
Time Frame: Baseline; Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 1 | 4
g/day | -0.177 | -2.151 (2.2591)

3. Secondary Outcome: Change From Baseline (Day 1) in Estimated Glomerular Filtration Rate (eGFR) at Week 16
Time Frame: Baseline; Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 1 | 4
mL/min/1.73 m^2 | -59.4 | -2.0 (11.35)

4. Secondary Outcome: Change From Baseline (Day 1) in Urine Protein Creatinine Ratio (UPCR) at Week 16
Description: UPCR was assessed by urine protein excretion during a 24-hour urine collection.
Time Frame: Baseline; Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 1 | 4
mg/mg | -4.407 | -0.808 (0.7539)

5. Secondary Outcome: Percentage of Participants With Partial Remission at Week 16
Description: Partial Remission was defined as urine protein excretion below < 3 g/day and urine protein excretion decrease by ≥ 50% among participants with baseline (Day 1) nephrotic range proteinuria [urine protein excretion ≥ 3 g/day]; or urine protein excretion decrease by ≥ 50% among participants with subnephrotic range proteinuria [urine protein excretion < 3 g/day]).
Time Frame: Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 1 | 4
percentage of participants | 0 | 50.0

6. Secondary Outcome: Percentage of Participants With Complete Remission at Week 16
Description: Complete Remission was defined as urine protein excretion below 0.5 g/day, with no hematuria.
Time Frame: Week 16
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Lanraplenib 30 mg | Filgotinib 200 mg
Number analyzed (Participants) | 1 | 4
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date plus 30 days (maximum: 56 weeks)
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Up to Week 16: Lanraplenib 30 mg: Participants received lanraplenib 30 mg tablet + filgotinib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase.
- Up to Week 16: Filgotinib 200 mg: Participants received filgotinib 200 mg tablet + lanraplenib placebo tablet orally once daily for 16 weeks in Blinded Treatment Phase.
- After Week 16: Lanraplenib 30 mg: At Week 16, participants who achieved ≥ 35% reduction in urinary protein excretion from baseline continued to receive same blinded study treatment (lanraplenib 30 mg tablet + filgotinib placebo tablet orally once daily) for additional 16 weeks.
  After 32 weeks of blinded treatment, participants who had ≥ 35% reduction in urinary protein excretion from baseline continued their assigned blinded treatment for additional 20 weeks in Extended Blinded Treatment Phase.
- After Week 16: Filgotinib 200 mg: At Week 16, participants who achieved ≥ 35% reduction in urinary protein excretion from baseline continued to receive same blinded study treatment (filgotinib 200 mg tablet + lanraplenib placebo tablet orally once daily) for additional 16 weeks.
  After 32 weeks of blinded treatment, participants who had ≥ 35% reduction in urinary protein excretion from baseline continued their assigned blinded treatment for additional 20 weeks in Extended Blinded Treatment Phase.
- After Week 16: Lanraplenib 30 mg to Filgotinib 200 mg: At Week 16, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from baseline to Week 16 switched treatment and received filgotinib 200 mg + lanraplenib placebo for additional 16 weeks.
  At Week 32, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from Week 16 to Week 32 could continue whichever treatment that led to the greatest reduction in urinary protein excretion, or either treatment per investigator's discretion for additional 20 weeks in Extended Blinded Treatment Phase.
- After Week 16: Filgotinib 200 mg to Lanraplenib 30 mg: At Week 16, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from baseline to Week 16 switched treatment and received lanraplenib 30 mg + filgotinib placebo for additional 16 weeks.
  At Week 32, participants who did not achieve a ≥ 35% reduction in urinary protein excretion from Week 16 to Week 32 could continue whichever treatment that led to the greatest reduction in urinary protein excretion, or either treatment per investigator's discretion for additional 20 weeks in Extended Blinded Treatment Phase.
Arm/Group | Up to Week 16: Lanraplenib 30 mg | Up to Week 16: Filgotinib 200 mg | After Week 16: Lanraplenib 30 mg | After Week 16: Filgotinib 200 mg | After Week 16: Lanraplenib 30 mg to Filgotinib 200 mg | After Week 16: Filgotinib 200 mg to Lanraplenib 30 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/0 | 0/3 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/5 | 0/0 | 0/3 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 3/5 | 0/0 | 1/3 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Up to Week 16: Lanraplenib 30 mg (N=4) | Up to Week 16: Filgotinib 200 mg (N=5) | After Week 16: Lanraplenib 30 mg (N=0) | After Week 16: Filgotinib 200 mg (N=3) | After Week 16: Lanraplenib 30 mg to Filgotinib 200 mg (N=1) | After Week 16: Filgotinib 200 mg to Lanraplenib 30 mg (N=1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Up to Week 16: Lanraplenib 30 mg (N=4) | Up to Week 16: Filgotinib 200 mg (N=5) | After Week 16: Lanraplenib 30 mg (N=0) | After Week 16: Filgotinib 200 mg (N=3) | After Week 16: Lanraplenib 30 mg to Filgotinib 200 mg (N=1) | After Week 16: Filgotinib 200 mg to Lanraplenib 30 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Gilead made a decision to discontinue enrollment after very low enrollment over 16 months. This decision was not due to any safety concerns. Only 9 participants were enrolled and 3 participants completed study, no inferential analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT03285711/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03285711/SAP_001.pdf